CLINICAL TRIAL: NCT06675825
Title: A Novel Endoscopic Attachment Cap for Benign Esophageal Stricture Dilation in Children: a Randomized, Multicentric Pilot Study.
Brief Title: An Innovative Endoscopic Cap for Dilating Benign Esophageal Strictures in Children
Acronym: BOUGIE-PED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Vasiliki Spyropoulou, Principal Investigator, University Children's Hospital, Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BASEC2023-D0111; SNCTP000005847 (Registry Identifier: Portal for clinical trials in Switzerland (SNCTP))
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Stenosis; Esophageal Dilation
Keywords: esophageal stricture; esophageal dilation; pediatric gastroenterology
MeSH Terms: conditions — Esophageal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group 1: BougieCap (Experimental): Patients randomized into this group will undergo the dilation using the BougieCap.
  Interventions: Device: BougieCap
- Study Group 2: Standard treatment (Active Comparator): Patients randomized to the standard treatment arm will be provided one of the two standard dilation techniques, Savary- Bougie dilation or balloon dilation. This procedure could take place under endoscopic or radiological control.
  Interventions: Device: Savary-Bougie (A) or balloon dilation (B)

INTERVENTIONS:
Device: BougieCap — The BougieCap is attached to the tip of the endoscope, offers direct visual and tactile control and the endoscope acts as a carrier of the radial and longitudinal force vectors for the dilation.
  Other Names: Esophageal dilation
  Arms: Study Group 1: BougieCap
Device: Savary-Bougie (A) or balloon dilation (B) — A: In the Savary- Bougie treatment, dilators of different sizes are advanced to dilate the stenosis. The same procedure is then repeated with the next larger dilator, with the position of the dilator being checked radiologically each time.
  B: In the case of balloon dilation, a balloon is inserted and inflated at the level of the stenosis. Depending on the age of the child and possibly also the etiology of the stenosis, different balloons sizes are applied, which are then maintained inflated for about one until three minutes and the respective pressure. This procedure could take place under endoscopic or radiological control.
  Other Names: Dilation of esophageal stricture; Esophageal dilation
  Arms: Study Group 2: Standard treatment

SUMMARY:
The goal of this study is to find out if using the BougieCap device is a safe and effective way to stretch narrow areas in the esophagus (food pipe) in children. The main questions this study wants to answer are:

* Does the BougieCap work well to treat narrow areas in the esophagus comparing with other methods to widen these narrow areas?
* Is BougieCap easy to use and does it cause fewer problems or discomfort for children?

Researchers will compare two groups: one using the BougieCap, and the other using traditional methods like balloon dilation, to see which one works better and is safer.

Participants will:

* Answer questions about their symptoms before treatment, 24 hours after, and 14 days later.
* Complete these questions during regular hospital visits or over the phone for the final check-up.

This study does not involve any extra risks or burdens for the participants.

DETAILED DESCRIPTION:
There are two categories of esophageal stricture in children: acquired and congenital. The development of benign esophageal stricture is based on significant fibromuscular alterations, inflammation in residual muscle layers and a deposition of collagen based on an inflammatory process . In children, these changes are most common in the context of a postoperative anastomotic stenosis in the case of esophageal atresia (usually type IIIb according to Vogt), as well as after caustic injury, peptic stricture and eosinophilic esophagitis. Rarely, children are born with congenital esophageal stricture. Therapeutic radiation can lead to stenoses requiring dilation. Likewise, children suffering from epidermolysis bullosa can suffer from esophageal stenosis. In rare cases, the ingestion of a foreign body in children causes symptomatic stenosis as a buried foreign body covered by esophageal hyper granulated tissue. Malignant stenosis is not considered in this study, as its treatment is different.

There are different options for endoscopic esophageal dilations of clinically relevant esophageal strictures, which promise effective treatment. Relevant strictures are usually noticed by dysphagia.

One possible dilation method uses the Savary-Gilliard bougies. These are wire-guided polyvinyl dilators. The advancement of the wire is performed under radiological fluoroscopy. Once the guide wire is placed into the stomach, the dilator is passed over the guidewire, lubricated, and pushed over the stenosis in order to dilate the stenotic area. There are also non-guidewire bougie dilators. Longitudinal shearing force and radial force occurs when the dilator passes across the stenotic area. Initially, the size of the dilator that corresponds to the diameter of the stenosis is used. The same procedure is then followed stepwise with a larger dilator of 1mm, respectively. It is generally recommended not to increase the dilator size more than 3mm in a single session.

A major disadvantage of this method is the exclusively tactile control of the dilation. At the end of the Bougie dilation, the result should be checked by reinserting the endoscope to rule out deeper mucosal injuries and persistent bleeding.

Furthermore, there is experience in the treatment of esophageal stenosis in children with balloon dilations. The balloon is inserted either blind or under endoscopic control, The balloon is then mostly inflated to 1 mm beyond the estimated stenosis diameter and the pressure is maintained for 1 minute or less. The dilation may be controlled radiologically or endoscopically. A dilation up to 5mm above the initial stricture diameter may not increase the risk of perforation. Only radial forces arise. Here, too, insufficient visual control is to be criticized. In particular, the distal area of the stenosis cannot be viewed during the procedure, or only with difficulty. In addition to the poor visual control, there is no tactile control of the dilation, since the volume of liquid applied to the balloon determines the diameter. Furthermore, there is no standard protocol for the stepwise dilation that is required for treating children at different ages. Finally, small esophageal balloons specifically for small children are missing, which is why balloon catheters from other areas and indications are used (e.g. urological balloon catheters, biliary catheters), respectively.

Due to the severely restricted visual control of the dilation with the current dilation techniques, a conical cap made of transparent plastic was developed that can be attached to the tip of standard endoscopes, the BougieCap (Ovesco, Tübingen). The cap is a single-use product, available in different outer diameters (7- 16mm) and offers direct visual and tactile control upon introduction into the upper gastrointestinal tract under visual and tactile control. The advantage of this technique is that the endoscope acts as a carrier of the radial and longitudinal force vectors for the dilation. A comparable technique is one with the optical dilator, a clear, over-the-scope bougie with sequential dilating segments. However, the limitation of this optical dilator is that it can only be used for the dilation of relatively large stenoses (from 15mm) due to the large diameter. A main reason why the optical dilator is not suitable for children.

There are currently no studies in the literature investigating the use of the BougieCap technique for treating benign esophageal strictures in children.

The aim of this randomized controlled pilot study is to demonstrate the probable efficacy of the BougieCap technique, the improvement of patient and operator dependent conditions and the absence or reduction of related adverse events such as perforations, bleeding, infections as well as the number of dilation sessions and intervals, compared to the above mentioned other techniques.

The BougieCap is an endoscopic attachment cap for bougienage/dilatation of stenoses and strictures of the upper gastrointestinal tract. No specific restrictions based on age, weight, health status or ethnicity. The decision on whether a patient is eligible for treatment with the product lies solely with the intended user. The BougieCap Ovesco is a medical device primarily composed of the cap and the adhesive tape that may come into contact with tissues (mainly Oesophagus mucosa) or bodily fluids (salive) during its application. As per regulatory standards, it's crucial to note that this device does not contain pharmaceuticals, human or animal tissues, their derivatives, or any other biologically active substances.

ELIGIBILITY:
Inclusion Criteria:

* Age under 18 years of age
* Indication for endoscopic esophageal dilation
* Benign stenosis
* Written Informed Consent signed by the subject and/or parent/legal representative (if applicable)

Exclusion Criteria:

* Stenosis that cannot be treated endoscopically
* Malignant esophageal strictures
* Contraindications and limitations of the MD as described in the instructions for use

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful dilation | Directly after the intervention
  Satisfactory dilation of the stenosis according to the operator

CONTACTS AND LOCATIONS:
Locations (3):
- Maternal and Child Health Department, University Hospital - Umberto I Sapienza - University of Rome,, Rome, Italy
- Switzerland (2):
  - University Children's Hospital Zurich, Zurich, Canton of Zurich
  - Universitäts-Kinderspital beider Basel, Basel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoepfer AM, Henchoz S, Biedermann L, Schreiner P, Greuter T, Reinhard A, Senn J, Franke A, Burri E, Juillerat P, Simon HU, Straumann A, Safroneeva E, Godat S. Technical feasibility, clinical effectiveness, and safety of esophageal stricture dilation using a novel endoscopic attachment cap in adults with eosinophilic esophagitis. Gastrointest Endosc. 2021 Nov;94(5):912-919.e2. doi: 10.1016/j.gie.2021.05.017. Epub 2021 May 15. PMID 34004192
- [Background] Lafeuille P, Yzet C, Bonniaud P, Rostain F, Ponchon T, Rivory J, Pioche M. Use of a bougie-shaped cap for dilation with direct visual control for an esophageal stricture induced by radiation therapy. Endoscopy. 2023 Dec;55(S 01):E18-E19. doi: 10.1055/a-1929-9317. Epub 2022 Sep 16. No abstract available. PMID 36113487
- [Background] Walter B, Schmidbaur S, Rahman I, Albers D, Schumacher B, Meining A. The BougieCap - a new method for endoscopic treatment of complex benign esophageal stenosis: results from a multicenter study. Endoscopy. 2019 Sep;51(9):866-870. doi: 10.1055/a-0959-1535. Epub 2019 Jul 23. PMID 31342473
- [Background] Ghiselli A, Bizzarri B, Ferrari D, Manzali E, Gaiani F, Fornaroli F, Nouvenne A, Di Mario F, De'Angelis GL. Endoscopic dilation in pediatric esophageal strictures: a literature review. Acta Biomed. 2018 Dec 17;89(8-S):27-32. doi: 10.23750/abm.v89i8-S.7862. PMID 30561414
- [Background] Dall'Oglio L, Caldaro T, Foschia F, Faraci S, Federici di Abriola G, Rea F, Romeo E, Torroni F, Angelino G, De Angelis P. Endoscopic management of esophageal stenosis in children: New and traditional treatments. World J Gastrointest Endosc. 2016 Feb 25;8(4):212-9. doi: 10.4253/wjge.v8.i4.212. PMID 26962403
- [Background] Jones MP, Bratten JR, McClave SA. The Optical Dilator: a clear, over-the-scope bougie with sequential dilating segments. Gastrointest Endosc. 2006 May;63(6):840-5. doi: 10.1016/j.gie.2005.08.042. PMID 16650550
- [Background] Clark SJ, Staffa SJ, Ngo PD, Yasuda JL, Zendejas B, Hamilton TE, Jennings RW, Manfredi MA. Rules Are Meant to Be Broken: Examining the "Rule of 3" for Esophageal Dilations in Pediatric Stricture Patients. J Pediatr Gastroenterol Nutr. 2020 Jul;71(1):e1-e5. doi: 10.1097/MPG.0000000000002687. PMID 32141993
- [Background] Cakmak M, Boybeyi O, Gollu G, Kucuk G, Bingol-Kologlu M, Yagmurlu A, Aktug T, Dindar H. Endoscopic balloon dilatation of benign esophageal strictures in childhood: a 15-year experience. Dis Esophagus. 2016 Feb-Mar;29(2):179-84. doi: 10.1111/dote.12305. Epub 2014 Dec 17. PMID 25515612
- [Background] Wallner O, Wallner B. Balloon dilation of benign esophageal rings or strictures: a randomized clinical trial comparing two different inflation times. Dis Esophagus. 2014 Feb-Mar;27(2):109-11. doi: 10.1111/dote.12080. Epub 2013 Apr 26. PMID 23621385
- [Background] Witzleben AV, Reiter R, Hoffmann T, Posovszky C. Buried Foreign Body in the Esophagus - Unusual Cause of Dysphagia in a 2-Year-Old Child. Klin Padiatr. 2019 Jul;231(4):214-216. doi: 10.1055/a-0942-1838. Epub 2019 Jun 17. No abstract available. PMID 31207651
- [Background] Shahein AR, Krasaelap A, Ng K, Bitton S, Khan M, Manfredi MA, Lerner DG. Esophageal Dilation in Children: A State of the Art Review. J Pediatr Gastroenterol Nutr. 2023 Jan 1;76(1):1-8. doi: 10.1097/MPG.0000000000003614. Epub 2022 Sep 19. PMID 36122370
- [Background] Collins MH, Alexander ES, Martin LJ, Grotjan TM, Mukkada VA, Sheil A, Abonia JP, Putnam PE, Rothenberg ME. Acquired Esophageal Strictures in Children: Morphometric and Immunohistochemical Analyses. Pediatr Dev Pathol. 2022 Mar-Apr;25(2):124-133. doi: 10.1177/10935266211041086. Epub 2021 Sep 13. PMID 34515576
- [Background] Standards of Practice Committee; Egan JV, Baron TH, Adler DG, Davila R, Faigel DO, Gan SL, Hirota WK, Leighton JA, Lichtenstein D, Qureshi WA, Rajan E, Shen B, Zuckerman MJ, VanGuilder T, Fanelli RD. Esophageal dilation. Gastrointest Endosc. 2006 May;63(6):755-60. doi: 10.1016/j.gie.2006.02.031. No abstract available. PMID 16650533